CLINICAL TRIAL: NCT04530097
Title: A Prospective, Double-blind, Randomized Controlled Study of Radiofrequency Ablation Combined With Melatonin in the Treatment of Stage IA NSCLC
Brief Title: Radiofrequency Ablation Combined With Melatonin in the Treatment of Stage IA NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ming Li, Associate senior doctor, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020KT128
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: NSCLC and Theropy
Keywords: NSCLC; radiofrequency ablation; Melatonin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RFA+MLT (Experimental): Radiofrequency ablation was performed immediately after enrollment, and melatonin treatment was given for 6 months after 1 week after radiofrequency.
  Interventions: Procedure: RFA
- RFA (No Intervention): Radiofrequency ablation was performed immediately after enrollment, and a placebo treatment program was given for 6 months after 1 week after radiofrequency.

INTERVENTIONS:
Procedure: RFA — Radiofrequency ablation was performed immediately after enrollment, and melatonin treatment was given for 6 months after 1 week after radiofrequency.
  Other Names: MLT
  Arms: RFA+MLT

SUMMARY:
Based on the recommendations of the guidelines, as well as the previous animal studies and clinical studies of our team, we designed and carried out prospective, randomized controlled, double-blind clinical studies to further expand the sample size to verify the efficacy of radiofrequency ablation combined with melatonin in the treatment of stage IA NSCLC. It is hoped that this combined treatment plan can delay the recurrence of lung cancer after RFA and prolong the survival time of patients.

DETAILED DESCRIPTION:
OBJECTIVES:

To verify the efficacy of radiofrequency ablation combined with melatonin in the treatment of stage IA non-small cell lung cancer, and explore new directions for the prevention and treatment of early stage non-small cell lung cancer.

OUTLINE:

This is a Prospective, double-blind, randomized controlled study. Using the same admission criteria, it is planned to enroll 260 patients, who will be randomly assigned 1:1. The experimental group: radiofrequency ablation combined with melatonin, and the control group: radiofrequency ablation combined with placebo.

Intervention group: Radiofrequency ablation was performed immediately after enrollment, and melatonin treatment was given for 6 months after 1 week after radiofrequency.

Control group: Radiofrequency ablation was performed immediately after enrollment, and a placebo treatment program was given for 6 months after 1 week after radiofrequency.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients can understand and voluntarily join this study, sign an informed consent form, and have good compliance.

  (2) Patients with peripheral early lung cancer who cannot tolerate surgery with poor cardiopulmonary function; (3) Patients with peripheral early-stage lung cancer who cannot tolerate surgery; (4) Patients with peripheral early lung cancer who are unwilling to undergo surgery; (5) The tumor is more than 1.0 cm away from large blood vessels or larger bronchi.

  (6) Age ≥18 years old and ≤85 years old; (7) ECOG PS score: 0-2 points; (8) Good coagulation function, platelet count ≥100×10^9/L, INR and PT≤1.5 times ULN; if the subject is receiving anticoagulation therapy, as long as the PT is within the intended use range of anticoagulation drugs; (9) Females of childbearing age should agree to use contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; serum or urine pregnancy test within 7 days before study entry Negative, and must be a non-lactating patient; men should agree to patients who must use contraception during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

* (1) Those with severe comorbidities, infection period, and immunocompromised persons; (2) Patients who are judged to seriously affect survival or cannot tolerate thoracoscopic surgery in pre-assessment; (3) Patients who have contraindications to radiofrequency ablation and cannot complete the treatment; (4) Merge other organ/system tumors. (5) At present, patients with long-term oral hormones and autoimmune diseases (6) Various bleeding diseases, acute infectious diseases, fever, women during pregnancy, (7) Recovery period after heart surgery or stent implantation. (8) Those who are difficult to cooperate to complete the baseline test; those who cannot take drugs regularly;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
overall survival rate，OS | 2 years
  From the beginning of randomization to the time of death due to any reason (patients who are lost to follow-up are the time of the last follow-up; patients who are still alive at the end of the study are the end of follow-up), when the survival curve reaches 2 years, the survival rate of patients.

SECONDARY OUTCOMES:
DFS | 2 years
  The time interval from the first medication to the observation of recurrence or metastasis, or death from any cause (calculated based on the previous event). Patients who have not relapsed, metastasized or died at the time of the data cutoff, and those who were lost to follow-up in the study will be counted on the date of their last tumor evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality, China